CLINICAL TRIAL: NCT03901105
Title: Evaluation of the Relationship Between Baseline Flortaucipir PET Signal and Cognitive Change in Subjects With Early Alzheimer's Disease Participating in the I8D-MC-AZES Protocol Addendum D5010C00009 (2.1) (Tau Imaging)
Brief Title: Evaluation of Flortaucipir PET Signal and Cognitive Change in Early Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-PX01
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Intervention Model Description: Physician PET scan readers are participants, blinded to demographic and clinical data from the source PET scans.
Masking Description: PET scans were obtained in an open-label fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flortaucipir PET Scan (Experimental): No study drug will be administered. Scans previously acquired from Study I8D-MC-AZES (NCT02245737, Eli Lilly and Company sponsor) will be read by independent, blinded readers.
  Interventions: Drug: flortaucipir F18; Procedure: Brain PET Scan

INTERVENTIONS:
Drug: flortaucipir F18 — No study drug will be administered. Scans previously acquired from Study I8D-MC-AZES (NCT02245737, Eli Lilly and Company sponsor) at baseline will be read by independent, blinded readers. IV injection, 240 megabecquerel (MBq) (6.5 mCi), single dose in AZES
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748
Procedure: Brain PET Scan — positron emission tomography (PET) scan of the brain

SUMMARY:
This study will evaluate whether visual interpretation of flortaucipir-PET (positron emission tomography) scans, examining patterns of tracer uptake at baseline, can predict the rate of clinically-meaningful cognitive decline due to AD after 18 months. All scans are acquired from cohorts of a previously completed study, I8D-MC-AZES (NCT02245737, lanabecestat, Eli Lilly and Company sponsor).

ELIGIBILITY:
Scan Reader Criteria (5 total readers):

* Board-certified in radiology or nuclear medicine
* Professional experience interpreting PET scans

Scan Criteria (205 total scans):

* Former enrollment in AZES Study
* Flortaucipir scan at baseline
* clinical dementia rating - sum of boxes (CDR-SB) assessment at 18 months

Scan Study Population (AZES Study):

* 55 to 85 years
* MCI due to AD or probable AD by National Institute on Aging-Alzheimer's Association criteria (Albert 2011
* mini-mental status exam (MMSE) of 20 to 30 inclusive
* CDR global score of 0.5 (MCI), or 0.5 or 1 (AD) with a memory box score ≥ 0.5, and a score of ≤85 on the Delayed Memory Index of the Repeatable Battery for the Assessment of Neuropsychological Status.
* Amyloid positive status confirmed by florbetapir PET or lumbar puncture

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Avid Radiopharmaceuticals
Locations (1):
- American College of Radiology, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu M, Pontecorvo MJ, Devous MD Sr, Arora AK, Galante N, McGeehan A, Devadanam C, Salloway SP, Doraiswamy PM, Curtis C, Truocchio SP, Flitter M, Locascio T, Devine M, Zimmer JA, Fleisher AS, Mintun MA; AVID Collaborators. Aggregated Tau Measured by Visual Interpretation of Flortaucipir Positron Emission Tomography and the Associated Risk of Clinical Progression of Mild Cognitive Impairment and Alzheimer Disease: Results From 2 Phase III Clinical Trials. JAMA Neurol. 2021 Apr 1;78(4):445-453. doi: 10.1001/jamaneurol.2020.5505. PMID 33587110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Scans were acquired from subjects previously enrolled in the AZES (NCT02245737) PET substudy (N=205), including mild AD (n=141) and mild cognitive impairment (MCI) due to AD (n=64).
Pre-assignment Details: To be included in the study, subjects had to have a valid baseline flortaucipir PET scan and clinical dementia rating (CDR) assessments at baseline and 18 months.
Groups:
- All Subjects: Mild AD and MCI due to AD from the flortaucipir PET scan arm
Period: Overall Study
Arm/Group | All Subjects
Started | 205
Completed | 205
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Scans: Mild AD and MCI due to AD from the flortaucipir PET scan arm
Arm/Group | All Scans
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 27
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 172
  More than one race | 0
  Unknown or Not Reported | 1
Flortaucipir PET Scan Result [Count of Participants; unit: Participants] — Majority read result of 5 independent readers. τAD++ (a pattern indicating spread of aggregated tau beyond the posterolateral temporal [PLT] lobe or occipital lobe); τAD+ (a pattern indicating aggregated tau confined to PLT and/or occipital lobe); or τAD- (inconsistent with an AD pattern).
  Participants
    tAD++ | 162
    tAD+ | 15
    tAD- | 28
Mean CDR-SB [Mean (Standard Deviation); unit: units on a scale] — Mean Clinical Dementia Rating - Sum of Boxes Score (CDR-SB). The CDR scale (Berg 1988) examines 6 cognitive functioning domains individually on a scale of 0 to 3. CDR Sum of Boxes is generated by summing the total score across domains. Scores range from 0 to 18, with higher scores indicating higher levels of cognitive impairment.
  units on a scale | 3.69 (1.475)

OUTCOME MEASURES:

1. Primary Outcome: Risk Ratio for AD Symptom Progression on CDR-SB
Description: Baseline flortaucipir F 18 PET imaging results were determined by majority read (see Baseline Characteristics for description). Clinically meaningful deterioration (CMD) was defined for the primary endpoint as a worsening of the Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) score of one point or more. The clinical dementia rating (CDR) examines 6 categories of cognitive functioning domains. Each domain is scored on a scale ranging from 0 to 3 (including 0.5). A CDR-SB was generated as the sum of the values in each of the 6 domains. The CDR-SB sum scores range from 0 to 18, with higher scores indicating greater cognitive impairment and a 1 point worsening is considered a clinically significant symptom change.
Time Frame: Within 18 months of scan
Measure: Count of Participants; unit: Participants
Groups:
- CMD (CDR-SB Change >=1): Subjects who experienced at least a 1 point worsening in CDR-SB score over 18 months
- No CMD: Subjects who experienced less than a 1 point worsening in CDR-SB score over 18 months
Arm/Group | CMD (CDR-SB Change >=1) | No CMD
Number analyzed (Participants) | 143 | 62
Participants
  tAD++ | 119 | 43
  tAD+ | 10 | 5
  tAD- | 14 | 14
Statistical Analysis 1: Comparison: CMD (CDR-SB Change >=1) vs No CMD; Scan results were grouped into τAD++ vs. non-τAD++ (τAD+ and τAD-) for the analysis; Test type: Other; p = 0.0313, log linear model — A priori threshold was two-sided 0.05; Adjusted for treatment arm (lanabecestat 20 mg, 50 mg, or placebo), baseline age, years of education (categorical), and baseline CDR-SB score; Risk Ratio (RR) = 1.36, 95% CI 2-sided [1.028 to 1.785] — τAD++ scans represent the numerator for risk, and τAD+/τAD- scans represent the denominator

2. Secondary Outcome: Risk Ratio for AD Symptom Progression on Various Clinical Measures
Description: Baseline flortaucipir F 18 PET imaging results were determined by majority read (see Baseline Characteristics for description). Clinically meaningful deterioration (CMD) was defined for the cognitive endpoints as follows: mini-mental status exam (MMSE) worsening of 3 points or greater, Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) worsening of 4 points or greater, Pfeffer's Functional Activities Questionnaire (FAQ) worsening of 3 points or greater, CDR global worsening of greater than 0 points. MMSE scores range from 0 to 30 with lower scores indicating worsening cognitive function. ADAS-Cog11 scores range from 0 to 70 with higher scores indicating worsening cognitive function. FAQ scores range from 0 to 30 with higher scores indicating worsening cognitive function. CDR global is scored on a 5 point scale (0, 0.5, 1, 2, 3) with higher scores indicating worsening cognitive function.
Time Frame: Within 18 months of scan
Population: All subjects were eligible for this analysis; however, row totals reflect subjects for whom clinical measure data was available at baseline and 18 months.
Measure: Count of Participants; unit: Participants
Groups:
- CMD Yes: Subjects who experienced CMD for the clinical measure as described above
- No CMD: Subjects who did not experience CMD for the clinical measure as described above
Arm/Group | CMD Yes | No CMD
Number analyzed (Participants) | 205 | 205
Participants
  MMSE: number analyzed (Participants) | 133 | 70
  MMSE: tAD++ | 112 | 49
  MMSE: tAD+ | 6 | 8
  MMSE: tAD- | 15 | 13
  ADAS-Cog: number analyzed (Participants) | 112 | 87
  ADAS-Cog: tAD++ | 98 | 59
  ADAS-Cog: tAD+ | 6 | 8
  ADAS-Cog: tAD- | 8 | 20
  FAQ: number analyzed (Participants) | 134 | 66
  FAQ: tAD++ | 111 | 47
  FAQ: tAD+ | 9 | 5
  FAQ: tAD- | 14 | 14
  CDR Global: number analyzed (Participants) | 87 | 118
  CDR Global: tAD++ | 71 | 91
  CDR Global: tAD+ | 7 | 8
  CDR Global: tAD- | 9 | 19
Statistical Analysis 1: Comparison: CMD Yes vs No CMD; Risk ratio for MMSE CMD. Scan results were grouped into τAD++ vs. non-τAD++ (τAD+ and τAD-) for the analysis; Test type: Other; p = .0833, log linear model — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for treatment arm (lanabecestat 20 mg, 50 mg, or placebo), baseline age, years of education (categorical), and baseline score; Risk Ratio (RR) = 1.35, 95% CI 2-sided [0.962 to 1.886] — τAD++ scans represent the numerator for risk, and τAD+/τAD- scans represent the denominator
Statistical Analysis 2: Comparison: CMD Yes vs No CMD; Risk ratio for ADAS-Cog11 CMD. Scan results were grouped into τAD++ vs. non-τAD++ (τAD+ and τAD-) for the analysis; Test type: Other; p = .0141, log linear model — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.77, 95% CI 2-sided [1.122 to 2.796] — τAD++ scans represent the numerator for risk, and τAD+/τAD- scans represent the denominator
Statistical Analysis 3: Comparison: CMD Yes vs No CMD; Risk ratio for FAQ CMD. Scan results were grouped into τAD++ vs. non-τAD++ (τAD+ and τAD-) for the analysis; Test type: Other; p = .0639, log linear model — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.32, 95% CI 2-sided [0.984 to 1.776] — τAD++ scans represent the numerator for risk, and τAD+/τAD- scans represent the denominator
Statistical Analysis 4: Comparison: CMD Yes vs No CMD; Risk ratio for CDR Global CMD. Scan results were grouped into τAD++ vs. non-τAD++ (τAD+ and τAD-) for the analysis; Test type: Other; p = .2814, log linear model — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.28, 95% CI 2-sided [0.815 to 2.020] — τAD++ scans represent the numerator for risk, and τAD+/τAD- scans represent the denominator

3. Secondary Outcome: Mean Change in Cognitive/Functional Assessments
Description: Mean change in cognitive/functional measures baseline between τAD++ and non-τAD++ (determined by baseline tau status), calculated by Mixed Model Repeat Measures (MMRM). CDR-SB scores range from 0 to 18, with higher scores indicating worsening cognitive impairment. MMSE scores range from 0 to 30 with lower scores indicating worsening cognitive function. ADAS-Cog11 scores range from 0 to 70 with higher scores indicating worsening cognitive function. FAQ scores range from 0 to 30 with higher scores indicating worsening cognitive function.
Time Frame: baseline and 18 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- τAD++ Scan Result: Subjects with a τAD++ scan result
- Non-τAD++ Scan Result: Subjects with a Non-τAD++ scan result
Arm/Group | τAD++ Scan Result | Non-τAD++ Scan Result
Number analyzed (Participants) | 162 | 43
units on a scale
  CDR-SB | 2.22 (0.215) | 1.31 (0.379)
  MMSE: number analyzed (Participants) | 161 | 42
  MMSE | -4.89 (0.377) | -2.12 (0.647)
  ADAS-Cog11: number analyzed (Participants) | 157 | 42
  ADAS-Cog11 | 6.53 (0.660) | 1.97 (1.181)
  FAQ: number analyzed (Participants) | 158 | 42
  FAQ | 5.22 (0.537) | 2.68 (0.895)
Statistical Analysis 1: Comparison: τAD++ Scan Result vs Non-τAD++ Scan Result; MMRM testing the difference between CDR-SB least squares mean changes of tAD++ and Non-tAD++ (tAD+ and tAD-). The unstructured covariance structure (UN) was used; Test type: Other; p = .0305, Mixed Models Analysis — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for baseline clinical score, age, years of education (categorical), and treatment arm (lanabecestat - 20mg or 50mg - or placebo)
Statistical Analysis 2: Comparison: τAD++ Scan Result vs Non-τAD++ Scan Result; MMRM testing the difference between MMSE least squares mean changes of tAD++ and Non-tAD++ (tAD+ and tAD-). The unstructured covariance structure (UN) was used; Test type: Other; p < 0.0001, Mixed Models Analysis — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: τAD++ Scan Result vs Non-τAD++ Scan Result; MMRM testing the difference between ADAS-Cog11 least squares mean changes of tAD++ and Non-tAD++ (tAD+ and tAD-). The unstructured covariance structure (UN) was used; Test type: Other; p = 0.0006, Mixed Models Analysis — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: τAD++ Scan Result vs Non-τAD++ Scan Result; MMRM testing the difference between FAQ least squares mean changes of tAD++ and Non-tAD++ (tAD+ and tAD-). The unstructured covariance structure (UN) was used; Test type: Other; p = 0.0097, Mixed Models Analysis — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Inter-Reader Reliability of Reader Interpretation of Flortaucipir F 18 PET Imaging
Description: As measured by Fleiss' Kappa across all scans read. Fleiss' kappa is a statistical measure for assessing the reliability of agreement between a fixed number of raters when assigning categorical ratings to a number of items or classifying items. Fleiss' kappa can range from -1 to 1 with 1 indicating perfect agreement between the readers. Read results binarized as τAD++ or non-τAD++.
Time Frame: baseline scan
Measure: Number (95% Confidence Interval); unit: kappa coefficient
Groups:
- All Subjects/All Readers: All subjects scans included in the study across 5 independent readers
Arm/Group | All Subjects/All Readers
Number analyzed (Participants) | 205
kappa coefficient | 0.754 [0.711 to 0.797]

ADVERSE EVENTS:
Time Frame: Not applicable, as no new patients received treatment as part of this study.
Description: Adverse event data were not collected in this study.
Groups:
- Single Arm, Randomly Sequenced Flortaucipir F18 Scans: No study drug was administered for this study. Scans were previously acquired from Study I8D-MC-AZES (NCT02245737, Eli Lilly and Company sponsor) and were read by five independent, blinded readers.
  Flortaucipir F18: No study drug was administered for this study.
Arm/Group | Single Arm, Randomly Sequenced Flortaucipir F18 Scans
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03901105/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03901105/SAP_001.pdf